CLINICAL TRIAL: NCT06259643
Title: Clinical and Psychosocial Impact of Power Wheelchair Soccer for Individuals Presenting With Physical Impairments
Brief Title: Effects of Power Wheelchair Soccer for Individuals Presenting With Physical Impairments
Acronym: chair-soccer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FOOT FAUTEUIL
Record Dates: First submitted 2024-01-23; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Neuromuscular Diseases; Cerebral Palsy
MeSH Terms: conditions — Neuromuscular Diseases; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Power wheelchair soccer (Experimental): soccer game performed with a wheelchair
  Interventions: Other: Power wheelchair soccer

INTERVENTIONS:
Other: Power wheelchair soccer — Participants will practice power wheelchair soccer during the course of the power wheelchair soccer season (starting in November 2023 and ending in June 2024). Sessions are given once a week, by a coach with experience in this adaptive sport.

SUMMARY:
This study is a prospective interventional study. It will be conducted at a single center with participants who have neuromotor impairments. The primary objective is to assess and measure the clinical and psychosocial effects of a season of power wheelchair soccer among its participants presenting with severe motor impairments due to neuromuscular lesion.

A maximum of twenty participants will be recruited and included in the same group. Data collection will be performed before, during, and after the wheelchair soccer season. The study will span the entire season, starting in November 2023 and ending in June 2024.

Clinical and psychosocial assessments will be conducted every 3 months. Each assessment session will last 2 hours per participant. Before and after the wheelchair soccer season matches, we will evaluate parameters related to the physical load of the sport. These evaluations will last 10 minutes per participant.

ELIGIBILITY:
Inclusion Criteria:

* Being a male or female between the ages of 12 and 50.
* Presenting with severe motor impairments due to neuromotor and/or musculoskeletal impairment.
* Using a power wheelchair in everyday life.
* Being part of a power wheelchair soccer team.
* Committing to participating in the 2023-2024 season of their sport within the team.

Exclusion Criteria:

* Practicing another adaptive sport outside of power wheelchair soccer in a regular way (once a week or more).
* Occasionally practicing power wheelchair soccer (twice a month or less).
* Presenting with severe cognitive impairments affecting understanding of instructions on how to answer questionnaires and undertake tests.
* Presenting with contraindications towards the practice of an adaptive sport such as power wheelchair soccer.

  * Participating in another study at baseline.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Balance | Throughout the entire study (an average of 8 months)
  Balance will be measured using the Trunk control measurement scale. Scores range from 0 to 58, where a higher score displays better trunk control.
Balance | Throughout the entire study (an average of 8 months)
  Balance will be measured using the Level of sitting scale. Levels range from 1 to 8, where a higher score demonstrates better sitting balance.
Balance | Throughout the entire study (an average of 8 months)
  Balance will be measured using the function section of the Seated Postural Control measure. Scores range from 12 to 48, where a higher score is attributed to individuals with better postural control.
Sensorimotor impairment | Throughout the entire study (an average of 8 months)
  Sensorimotor impairment will be measured by the Fugl-Meyer assessment.
Hyperactivity of the muscles | Throughout the entire study (an average of 8 months)
  Hyperactivity of the muscles will be measured using the Australian Spasticity Assessment scale of the upper-limb main muscle groups. Scores per muscle groups range from 0 to 4, where a higher score represents greater spasticity and more hyperactivity in the muscle group.
Hyperactivity of the muscles | Throughout the entire study (an average of 8 months)
  Hyperactivity of the muscles will be measured using the Penn Spasm Frequency Scale. Scores range from 0 to 4, where a higher score represents more frequent spasms and hyperactivity of the muscles.
Pain | Throughout the entire study (an average of 8 months)
  Pain perceived by the participants in their daily life will be measured using the PROMIS pain-pediatric Short Form V2 questionnaire. Scores range from 8 to 40, where a higher score displays more pain in everyday life.
Quality of life | Throughout the entire study (an average of 8 months)
  Quality of life will be assessed using the KIDSCREEN 27 questionnaire. Scores range from 10 and 50, where 50 represents a very high health-related quality of life.
Skills to manage and move power wheelchair | Throughout the entire study (an average of 8 months)
  Skills to manage and move power wheelchair will be assessed by the Wheelchair Skills Test Questionnaire version 4.2. Scores range from 0 to 100%, where a greater percentage represents better skills.
Social participation | Throughout the entire study (an average of 8 months)
  Social participation will be assessed using the Questionnaire of young people's participation.Scores range from 0 to 239, where a higher score displays greater social participation.
Autonomy during activities of daily life | Throughout the entire study (an average of 8 months)
  Autonomy during activities of daily life will be assessed using the Impact on participation and autonomy questionnaire. A participation score (range: 30-155) and a problem score (0-16) are produced by summing items in each scale. For both, a higher score represent poorer autonomy and more severe difficulty.
Strength of the upper-limbs | Throughout the entire study (an average of 8 months)
  Strength of the main muscle groups of the upper-limb will be measured using a Microfet 2 dynamometer.
Passive range of motion the upper-limbs | Throughout the entire study (an average of 8 months)
  Passive range of motion of the upper-limbs will be measured using a goniometer.

SECONDARY OUTCOMES:
Body temperature | Throughout the entire study (an average of 8 months)
  Body temperature will be evaluated using a tympanic thermometer.
Blood oxygen saturation | Throughout the entire study (an average of 8 months)
  Blood oxygen saturation will be evaluated using a pulse oximeter.
Heart beat rate | Throughout the entire study (an average of 8 months)
  Heart beat rate will be evaluated using a heart rate monitor.
Blood pressure | Throughout the entire study (an average of 8 months)
  Blood pressure will be evaluated on the left upper-arm with a tensiometer. Both systolic and diastolic pressure will be recorded.

OTHER OUTCOMES:
Satisfaction with the power wheelchair soccer practices | Throughout the entire study (an average of 8 months)
  Satisfaction with the power wheelchair soccer practices will be evaluated on a 10 point Likert-scale. A higher score displays greater satisfaction with the practices.
Demographic variables | Throughout the entire study (an average of 8 months)
  Participants' age, sex, origin of physical impairment, motor impairment severity, hours of physical therapy per week, as well as motor impairment severity, will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromusculoskeletal Lab, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No